CLINICAL TRIAL: NCT00207961
Title: The Threshold Value of Regional Cerebral Oxygenation in Detecting Cerebral Ischemia
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR-93-43
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-09

CONDITIONS: Cerebral Ischemia; Regional Cerebral Oxygenation
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Using patients receiving spinal anesthesia as a model to evaluate the treshold value of cerebral oximeter to detect the symptoms of cerebral ischemia

DETAILED DESCRIPTION:
56 patients has been recruited for the analysis of relationship between the symptoms of cerebral ischemia and the value of cerebral oximeter. All patients were recieved spinal anesthesia for the procedure of Ceserean section.

ELIGIBILITY:
Inclusion Criteria: patients who are going to undergo Cesarean section under spinal anesthesia

Exclusion Criteria: conditons contraindicated for regional anesthesia

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Dates: Start 2003-10; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Hung C Cheng, M.D., Study Director — Anesthetic Department
Locations (1):
- Anesthetic Department, Taichung, Taiwan